CLINICAL TRIAL: NCT06949397
Title: Effect Of Menstrual Belt And Stress Ball Application On Pain Intensity In Women With Dysmenorrhea
Brief Title: The Effect of the Menstrual Belt Stress Ball on Pain in Women With Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gedik University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GEDIKU-EBE-ME-01
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Education
Keywords: pain; dismenore; Menstruation belt; stress ball
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Menstrual belt group (Experimental): Before any procedure was performed, the women included in the Experiment 1 group were administered the Volunteer Information and Consent Form, Introductory Information Form, Visual Pain Scale, Dysmenorrhea Impact Scale-Revised Short Form (DIS-R), and Menstruation Symptom Scale when they complained of dysmenorrhea during menstruation. In participants with dysmenorrhea pain of 4 or more, the electric menstrual belt that applies hot massage was used to all participants in a way that it did not come into direct contact with the skin over the top of the clothes during the 20 minutes planned for women to relieve pain on the day of menstruation. After the application was over, the participant was asked to fill out the Visual Pain Scale (VAS) form again to evaluate the effect of the use of the menstrual belt on the dysmenorrhea complaint felt during menstruation.
  Interventions: Other: Change in VAS voice performance score following the characteristics of the menstrual cycle of two women
- Stress Relief Ball group (Experimental): The women included in the Experimental 2 group were administered the Volunteer Information and Consent Form, Introductory Information Form, Visual Pain Scale, Dysmenorrhea Impact Scale-Revised Short Form (DERS-R), and Menstruation Symptom Scale when they complained of dysmenorrhea during menstruation before any procedure was performed. At this stage, dysmenorrhea complaint was given to the participant with a score of 4 and above. On the day of menstruation, when dysmenorrhea complaint started, the women were given the anti-stress soft ball toy to squeeze in their hands within the planned 20 minutes. After the application was over, the participant was asked to fill out the Visual Pain Scale (VAS) form again to evaluate the effect of the use of anti-stress soft ball on the dysmenorrhea complaint experienced during menstruation.
  Interventions: Other: Change in VAS voice performance score following the characteristics of the menstrual cycle of two women
- Control group (No Intervention): Women enrolled in the control group did not undergo any procedure, and before and after the procedure, the informed consent form, the introductory information form, the visual pain scale, the Dysmenorrhea Impact Scale-Revised Short Form (DIS-R), and the menstrual symptom scale were used. Women with a Dysmenorrhea Impact Score of 4 and above were monitored for 20 minutes without intervention by starting a stopwatch on the telephone. At the end of the 20-minute follow-up period given to the control group, the stopwatch on the phone was stopped. The control group was asked to fill out the Visual Pain Scale (VAS) form again to evaluate the dysmenorrhea complaint scores after the follow-up was over. After answering the questions in the data collection forms, the individual questions were answered.

INTERVENTIONS:
Other: Change in VAS voice performance score following the characteristics of the menstrual cycle of two women — application of menstrual belt and stress ball to women in the research group
  Other Names: studying the effect of the stress ball
  Arms: Menstrual belt group; Stress Relief Ball group

SUMMARY:
This study will be conducted as a randomized controlled quasi-experimental study to determine the effect of hot massage menstrual belt and stress relief ball application on pain intensity in women with dysmenorrhea. The study will include 105 women with dysmenorrhea (midwife, nurse, doctor, cleaning staff, secretary) who meet the inclusion criteria. Female participants between the ages of 18-45 will be randomly divided into three groups as experimental group 1 (n=35), experimental group 2 (n=35) and control group (n=35) by envelope method. Data will be collected using Informed Consent Form, Descriptive Information Form, Visual Pain Scale (VAS), Dysmenorrhea Impact Scale-Revised Short Form (DIS-R) and Menstrual Symptoms Scale. Descriptive Information Form, Visual Pain Scale (VAS), Dysmenorrhea Impact Scale-Revised Short Form (DIS-R) and Menstrual Symptom Scale will be applied to the three groups before the application. During the application, experimental group 1 will be given a menstrual belt with electric waist heating and vibration for 20 minutes. Experimental group 2 will be given a stress-relieving squeezing ball to feel its soft structure for the same period of time.The third group was determined as the control group and no application will be made. After the application, the participants will be asked to rate their pain intensity using the Visual Pain Scale (VAS) and record their pain scores.

DETAILED DESCRIPTION:
Menstruation is a physiological condition that significantly affects women's lives and is a process that recurs every month and is defined as bleeding that is expelled by periodic shedding of the endometrium layer in fertile females. The process of menstruation, which affects the lives of women of reproductive age, causes periodic monthly changes in the uterus and ovaries. These changes occur under the influence of hormones such as luteinizing hormone (LH), estrogen, follicle-stimulating hormone (FSH) and progesterone. The menstrual cycle is responsible for ovum production and prepares the uterus for pregnancy. The average length of the cycle is 28 days (ranging from 21-35 days), and the cycle is recognized as one that begins in a woman's life at menarche and continues until menopause.Pain during menstruation is characterized by painful cramps usually on the first or second day of menstruation and is defined as dysmenorrhea. It is usually categorized into two types: primary and secondary. Primary dysmenorrhea is recurrent, cramping abdominal pain that occurs during menstruation without any identifiable pelvic pathology.Secondary dysmenorrhea occurs due to pelvic or uterine pathology (such as fibroids, endometriosis, infection, uterine and ovarian cysts and tumors).Secondary dysmenorrhea can begin at any time after menarche, but it can also present as a new symptom when a woman is in her 30s and 40s after the onset of the underlying condition.

The pain in dysmenorrhea usually starts in the first 1-2 years after menarche. The incidence of dysmenorrhea may vary because most women with this problem do not apply to any health institution. When we look at the researches, it has been found that approximately 25-90% of women in the reproductive period complain of dysmenorrhea. In dysmenorrhea, cramp-like pain, which is predominant in the suprapubic region, can sometimes be accompanied by various systemic symptoms such as nausea, vomiting, fatigue, irritability, changes in appetite, insomnia, diarrhea and headache.These symptoms can be experienced in different severities and can lead to significant medical and psychosocial problems.Dysmenorrhea reduces the quality of life of women by causing changes in their physical activities and social roles. By affecting daily activity and performance, it causes loss of working days, especially in working women, and absenteeism in women who are studying.Methods that can be used to prevent or reduce dysmenorrhea complaints; Hot treatment, Exercise, Transcutaneous electrical nerve stimulation (TENS), Vitamins, Acupuncture, distraction, menstrual belt can be recommended. In order to ensure effective coping with symptoms during menstruation, women should be educated, informed and behavior change should be ensured rather than drug treatment.

In our study, as a result of the literature review, there was no study on the hot massage electric waist-heated menstrual belt and stress ball squeezing, which are among the methods that can be used to prevent or reduce complaints in women with dysmenorrhea complaints. This study was planned to determine the effect of distraction with menstrual belt and stress relieving ball on women's pain intensity level during the menstrual cycle.

Methods:

In this study; It will be carried out as a randomized controlled quasi-experimental study to determine the effect of menstrual belt and stress relief ball application on pain intensity in women aged 18-45 years with dysmenorrhea.

Menstruation Symptom Scale permission to use the scale will be obtained by e-mail. In the Turkish validity and reliability article of Dysmenorrhea Impact Scale-Revised Short Form permission will be obtained for the measurement tool with the condition of citing the source. Ethics committee approval will be obtained by applying to Istanbul Gedik University Ethics Committee. After the ethics committee approval is obtained, a study permit will be obtained from the Istanbul Provincial Directorate of Health to conduct the research in Sultanbeyli State Hospital.

The data obtained in the study were analyzed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Number, percentage, mean and standard deviation were used as descriptive statistical methods in the evaluation of the data. Differences between the rates of categorical variables in independent groups were analyzed with Chi-Square tests.

Kurtosis and Skewness values were analyzed to determine whether the research variables were normally distributed. According to the relevant literature, kurtosis and skewness values between +1.5 and -1.5 (Tabachnick & Fidell, 2013) or +2.0 and -2.0 (George & Mallery, 2010) are accepted as an indicator of normal distribution. According to the results of the analysis, the kurtosis value for the total dysmenorrhea impact score was 0.605 and the skewness value was 0.589; the kurtosis value for the cognitive/emotional sub-dimension was 0.301 and the skewness value was 0.548; the kurtosis value for the physiological sub-dimension was 1.223 and the skewness value was 0.849. The kurtosis value for the total menstruation symptom score was 0.093 and the skewness value was 0.303; the kurtosis value for the negative effects sub-dimension was 0.128 and the skewness value was 0.281; the kurtosis value for the menstrual pain sub-dimension was 0.094 and the skewness value was 0.688; the kurtosis value for the coping methods sub-dimension was 1.047 and the skewness value was 0.049. These values indicate that all variables fit the normal distribution.In the analysis of the data, parametric.

Procedures:

The women who agreed to participate in the study and who met the sampling criteria were given verbal and written information about the study. The women who agreed to participate in the study were firstly informed about the purpose of the study, that permission was obtained from the hospital management and ethics committee to conduct the study, that their identity information was required for research consent, and that their identity information would be kept confidential by the researcher. A whatsapp group was established in order to learn more easily that women with dysmenorrhea working in the hospital had pain during menstruation and to reach them. After verbal and written consent was obtained from the women, it was determined which group they would be in by randomization. For randomization (35 people experiment 1, 35 people experiment 2, 35 people control group), the groups were determined by the envelope selection method in which the groups were written on the papers and the participants were distributed to experiment 1, experiment 2 or control group according to the paper they drew. In the application phase of the study, out of a total of 5 people who did not meet the inclusion criteria among the answers to the questions given in the pre-application questionnaire, 1 person with a chronic illness, 1 person with a psychological disorder, and 3 people with a visual pain scale (VAS) score below 4 were excluded from the study.

Instruments:

* Descriptive Information Form: It will be used to evaluate the participants' sociodemographic data and menstruation-related data. In order to determine the socio-demographic and general health-related characteristics, participants will be asked about group information, age, height, body mass index, marital status, education level, telephone number, e-mail address, occupation, smoking habit, exercise habit, general health status, psychiatric disease status. In order to determine the characteristics related to menstruation, participants will be asked about the type of menstruation, duration of menstrual discharge, number of pads per day, frequency of changing pads per day, age at first menstruation, period of menstruation, the day menstrual pain started, duration, pattern, the time when the pain was the most severe, the complaint of pain in her mother or siblings, the effect of pain on daily activities, the need to use medication, the time of taking medication, how many medications she used and the method she used other than medication to cope with pain.
* Visual Analog Scale (VAS): The Visual Analog Scale (VAS) was developed to determine the severity of pain in individuals. VAS is a safe, easily applicable measurement tool that is used to convert some values that cannot be measured numerically into numerical form and has been generally accepted in the world literature for many years. The VAS consists of a 10 cm long line with subjective descriptive statements at both ends of the scale (0 cm = no pain and 10 cm = excruciating pain). The individual places a mark on this 10 cm line in the appropriate place for his/her pain. A low score on the VAS indicates that the pain intensity of the individual is low or mild, while a high score indicates that the pain intensity is high or severe.
* Dysmenorrhea Impact Scale-Revised Short Form (DEÖ-R): The measurement tool developed by Gün Kakaşçı and Demirci in 2023 consists of 13 items and 2 sub-dimensions. The first 8 items are cognitive/emotional and the last 5 items are physiological sub-dimensions. There are no reverse items in the scale. The scale is a five-point Likert-type scale and is scored as Strongly Disagree (1), Disagree (2), Undecided (3), Agree (4), Strongly Agree (5). The higher the participants' scores on the scale, the higher their level of being affected by dysmenorrhea. The Cronbach's alpha value of the scale is 0.83. This measurement tool can be used especially in those who experience symptoms of primary dysmenorrhea
* Menstruation Symptom Scale (MSS): The Menstrual Symptom Scale (MSS) was developed in English by Chesney and Tasto in 1975 to assess menstrual pain and symptoms. It is a widely used scale in the United States and many other countries. In 2009, it was updated by Negriff et al. by re-evaluating its factor structure and usability in adolescents. The scale was adapted into Turkish by Güvenç et al. in 2014. Participants are asked to assign a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. The scale items were numbered according to the factors allocated for ease of use. Items 1-13 belong to the "Negative effects/somatic complaints" subscale, items 14-19 belong to the "Menstrual pain symptoms" subscale and items 20-22 belong to the "Coping methods" subscale. Cronbach's Alpha value is 0.86. It is a five-point Likert-type scale consisting of 22 items. The score obtained from the sub-dimensions is calculated by averaging the total score of the items in the sub-dimensions. An increase in the mean score for the sub-dimensions indicates an increase in the severity of menstrual symptoms related to that sub-dimension.

In the pre-application phase, the feasibility of the data collection forms and the experimental design were evaluated. In order to allocate volunteers to the experimental and control groups and to avoid negative results related to the experiment, the pre-application phase of the research was conducted on 10 people before the start of the research, and these people were not included in the research.

As there was no negative situation in the pre-application phase, the implementation phase of the research was started.

After the pre-application phase, the implementation phase began. Women who agreed to participate in the study were given verbal and written information about the study to those who met the sampling criteria. The women who agreed to participate in the study were first informed about the purpose of the study, that permission to conduct the research had been obtained from the hospital management and the ethics committee, that their identity information was required for research consent, and that their identity information would be kept confidential by the researcher. A Whatsapp group was created to make it easier to know and reach out to women with dysmenorrhea working in the hospital. After obtaining verbal and written consent from the women, randomization was used to determine which group they would be in. For the randomization (35 people in Experiment 1, 35 people in Experiment 2, 35 people in the control group), the groups were determined by the envelope selection method in which the groups were written on the papers and the participants were distributed to Experiment 1, Experiment 2 or the control group according to the paper they drew. Application phase of the research

ELIGIBILITY:
Inclusion Criteria:

* Not being pregnant
* Being a woman between the ages of 18-45
* Duration of the menstrual cycle being 1-7 days
* Duration of the menstrual cycle being between 26-30 days
* Complaint of pain during the menstrual period
* Not having entered menopause
* Having the symptom of dysmenorrhea
* Not having any systemic disease
* Read- being an author
* being able to communicate in Turkish
* being willing to participate in the study
* not using drugs containing analgesics during the mentrual cycle
* giving 4 points or more (severe pain) to mentruation pain out of 10 points on the VAS Visual Pain Scale

Exclusion Criteria:

* Being pregnant
* Having entered menopause
* Having no pain problems during the mentrual cycle
* Mentrual cycle duration lasting from 26 to more than 30 days
* Mentrual day being less than 3 and more than 7
* Having any systemic disease
* Using drugs containing analgesics during the mentrual cycle
* Using psychotherapeutic drugs
* Having secondary dysmenorrhea
* Giving mentrational pain 3 points or less (severe pain) out of 10 points on the VAS Visual Pain Scale

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 105 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
change in the vas visual pain scale of the research group after using the menstrual belt | 20 minutes after applying the menstrual belt and stress ball
  Women in the research group applied menstrual belt and stress ball

CONTACTS AND LOCATIONS:
Overall Officials: Melek ERDOĞDU, Principal Investigator — Gedik University School of Nursing İstanbul, Turkey
Locations (1):
- Gedik University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Güvenç, G., Seven, M., & Akyüz, A. (2014). Menstrüasyon Semptom Ölçeği'nin Türkçe'ye Uyarlanması. TAF Preventive Medicine Bulletin, 13(5).
- [Background] Gün Kakaşçı, Ç., & Coşkuner Potur, D. İ. L. E. K. (2022). Menstruation Impact Scale Development. Medical records-international medical journal (Online), 4(3).
- [Background] Güvey, H. (2019). Adölesanlarda primer dismenore ve tedavi tedavileri. Jinekoloji-Obstetrik ve Neonatoloji Tıp Dergisi, 16 (3), 160-166
- [Background] Gün, Ç. (2014). Dismenore etkilenmişlik ölçeğinin geliştirilmesi (Doctoral dissertation, Doktora Tezi, İstanbul).
- [Background] Boztaş Elverişli, G. (2022). Primer dismenoreli kadınlarda farmakolojik ve non-farmakolojik tedavinin etkinliğinin karşılaştırılması.
- [Background] Yürekdeler Şahin, N. (2017). Yüksek frekanslı TENS ile konnektif doku manipulasyonunun primer dismenore üzerine etkilerinin karşılaştırılması.
- [Background] Şaşmaz, Y. (2022). Çevrimiçi yoga temelli egzersiz programının primer dismenoreli kadınlarda etkisinin araştırılması (Master's thesis, İstanbul Medipol Üniversitesi, Sağlık Bilimleri Enstitüsü).
- [Background] Potur DC, Bilgin NC, Komurcu N. Prevalence of dysmenorrhea in university students in Turkey: effect on daily activities and evaluation of different pain management methods. Pain Manag Nurs. 2014 Dec;15(4):768-77. doi: 10.1016/j.pmn.2013.07.012. Epub 2013 Nov 11. PMID 24230963
- [Background] Potur, D. C. (2009). Lokal düşük Doz ısı uygulamasının Dismenore üzerine Etkileri (Doctoral dissertation, Marmara Universitesi (Turkey)).